CLINICAL TRIAL: NCT00346151
Title: The Safety and Efficacy of Belatacept, Antithymocyte Globulin, and Sirolimus in Recipients of Non-HLA-identical Living-donor Renal Transplants (ITN023ST)
Brief Title: Belatacept to Prevent Organ Rejection in Kidney Transplant Patients
Acronym: BESTT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopping rule-acute rejection threshold-was met based on local biopsy results
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN023ST
Record Dates: First submitted 2006-06-27; First posted 2006-06-29 (Estimated); Results first posted 2011-11-07 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Renal Transplant
Keywords: renal transplantation; kidney transplantation; renal allograft recipient; anti-rejection drugs; immunosuppression protocol; immunosuppression withdrawal
MeSH Terms: interventions — Abatacept; Sirolimus; Antilymphocyte Serum; thymoglobulin; Methylprednisolone; Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Belatacept (Experimental): Immunosuppressive protocol consisting of belatacept, glucocorticoids, antithymocyte globulin (ATG), and sirolimus.
  Interventions: Drug: Belatacept; Drug: Sirolimus; Drug: Anti-thymocyte globulin; Drug: methylprednisolone

INTERVENTIONS:
Drug: Belatacept — 10 mg/kg given intravenously (IV) on transplant (day 1), day 5, and at weeks 2, 4, 8 and 12, then 5 mg/kg IV every 4 weeks
  Other Names: LEA29Y; Nulojix
Drug: Sirolimus — 4 mg/day (oral tablet) at transplant (day 1), then dose adjusted to maintain serum trough level of 8-12 ng/mL for at least 1 year
  Other Names: Rapamycin; Rapamune
Drug: Anti-thymocyte globulin — 1.5 mg/kg given IV daily on days 1 through 4. Subjects are premedicated with glucocorticoids, acetaminophen 650 mg by mouth, and diphenhydramine 25- 50 mg by mouth prior to each dose.
  Other Names: ATG; anti-thymocyte immunoglobulin; Thymoglobulin®
Drug: methylprednisolone — 500 mg given IV at transplant (day 1), then given 250 mg IV on day 2 and given 0.5 mg/kg IV or prednisone 0.5 mg/kg given by mouth on days 3 and 4
  Other Names: Medrol; glucocorticoid

SUMMARY:
Belatacept is an experimental medication shown in clinical trials to have immune system suppression properties in people who have had renal (e.g., kidney) transplants. This study will determine whether a combination of anti-rejection drugs, including belatacept, can prevent the rejection of a first-time, non-human leukocyte antigen (HLA) identical renal transplant and allow patients to be safely withdrawn from anti-rejection therapy one year post-transplant.

DETAILED DESCRIPTION:
Drugs that suppress the immune system have contributed to increased success of transplantation; however, to prevent organ rejection, transplant recipients need to take immunosuppressive drugs for the rest of their lives. These drugs make patients more susceptible to infection and certain kinds of cancer. Belatacept is an experimental medication that specifically targets immune reactions against transplanted organs and has been shown to be effective in preventing kidney transplant rejection in previous clinical trials. Both thymoglobulin, an antibody, and sirolimus, an anti-rejection drug, prevent rejection by lowering the response of the immune system to the transplanted organ. This study will evaluate whether belatacept, along with thymoglobulin and sirolimus, is safe in kidney transplant patients. The study will also evaluate this regimen's potential to allow tapering and eventual discontinuation of all immunosuppressive drugs.

This study will last up to 4 years. At the time of transplant, participants will begin an immunosuppressive treatment regimen consisting of thymoglobulin, sirolimus, and belatacept. Participants will receive infusions of thymoglobulin on days 1 through 4, and a combination of oral sirolimus (daily) and belatacept infusions at day 5, then weeks 2, 4, 8, and monthly for at least 2 years. Dose reduction of belatacept will occur at 12 weeks post-transplant. At Year 2, eligible participants may choose to begin drug withdrawal or continue study therapy through the end of the study. Study visits will occur weekly for the first two months, then monthly. These visits will include belatacept treatment, general medical assessments, blood and urine collection, and other assessments to determine overall health of the recipient's immune system and kidney transplant and to better understand the way the immune system works in the acceptance or rejection of organ transplants.

*** IMPORTANT NOTICE: *** The National Institute of Allergy and Infectious Diseases and the Immune Tolerance Network do not recommend the discontinuation of immunosuppressive therapy for recipients of cell, organ, or tissue transplants outside of physician-directed, controlled clinical studies. Discontinuation of prescribed immunosuppressive therapy can result in serious health consequences and should only be performed in certain rare circumstances, upon the recommendation and with the guidance of your health care provider.

ELIGIBILITY:
Inclusion Criteria:

* Receiving first renal (e.g., kidney) transplant
* Transplant is from a non-HLA-identical living donor
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* Positive for anti-human globulin (AHG) or T-cell cross-match with the donor
* Receiving multiple-organ transplant
* History of cancer within the 5 years prior to study entry. Patients who have certain nonmelanoma skin cancers are not excluded
* Human immunodeficiency virus (HIV) infected
* Hepatitis B (HBV) or C (HCV) virus infected
* Other active infections
* Active tuberculosis (TB) infection within the 3 years prior to study entry
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Vincenti, MD, Principal Investigator — University of California, San Francisco; Christian Larsen, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Data access is provided to the public in Participant level data and additional relevant materials are available to the public in : 1.) the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts that also provides data analysis tools available to researchers; and 2.) TrialShare, the Immune Tolerance Network (ITN) Clinical Trials Research Portal that makes data from the consortium's clinical trials publicly available.

REFERENCES:
- [Background] Vincenti F, Larsen C, Durrbach A, Wekerle T, Nashan B, Blancho G, Lang P, Grinyo J, Halloran PF, Solez K, Hagerty D, Levy E, Zhou W, Natarajan K, Charpentier B; Belatacept Study Group. Costimulation blockade with belatacept in renal transplantation. N Engl J Med. 2005 Aug 25;353(8):770-81. doi: 10.1056/NEJMoa050085. PMID 16120857
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network (ITN) website — http://www.immunetolerance.org
- Available data/document: Individual Participant Data Set: SDY674 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY674 — ImmPort study identifier is SDY674
- Available data/document: Study Protocol: SDY674 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY674 — ImmPort study identifier is SDY674. The study protocol is available in the Design tab section.
- Available data/document: Study summary, -design, -synopsis,- medications, -demographics, -lab tests, -files: SDY674 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY674 — ImmPort study identifier is SDY674
- Available data/document: Individual Participant Data Set: ITN023ST — http://www.itntrialshare.org/project/Studies/ITN023STPUBLIC/Study%20Data/begin.view? — TrialShare is a clinical trials research portal developed by the Immune Tolerance Network (ITN) that makes data from the consortium's clinical trials publicly available.
- Available data/document: Protocol synopsis, -data and reports, -specimens availability: ITN023ST — http://www.itntrialshare.org/project/Studies/ITN023STPUBLIC/Study%20Data/begin.view? — TrialShare is a clinical trials research portal developed by the Immune Tolerance Network (ITN) that makes data from the consortium's clinical trials publicly available.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two centers in the United States enrolled five recipients of non-human leukocyte antigen (HLA)-identical living-donor-related renal transplants between January 2007 and January 2009.
Pre-assignment Details: At a screening visit, participants underwent procedures to establish inclusion/exclusion criteria and sign the informed consent form.
Period: Overall Study
Arm/Group | Belatacept
Started | 5
Completed | 2
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Groups:
- Immunosuppression Withdrawal: Daclizumab, antithymocyte globulin, sirolimus, or belatacept dosing with the intention of immunosuppression withdrawal
Arm/Group | Immunosuppression Withdrawal
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Acute Rejection at 6-Months
Description: Cumulative incidence of acute rejection[1] at 6 months post-transplant based on local pathology biopsy reads
  1. Diagnosis of acute rejection was made by renal (kidney) biopsy using the Banff 97 criteria. The Banff 97 diagnostic category for renal allograft biopsies is an international standardized histopathological classification. Acute rejection is defined by a renal biopsy demonstrating a Banff 97 classification of Grade IA or greater[2]
  2. Reference: Racusen LC, Solez K, Colvin RB et al,The Banff 97 working classification of renal allograft pathology. Kidney Int,55: 713-723, 1999
Time Frame: 6 months post-transplant
Population: Intent to Treat
Measure: Number; unit: Participants
Arm/Group | Immunosuppression Withdrawal
Number analyzed (Participants) | 5
Participants | 3
Statistical Analysis 1: Comparison: Immunosuppression Withdrawal; Proportion of participant's cumulative incidence of acute rejection at 24 weeks with 95% exact binomial confidence interval. Local biopsy reads were used in determining primary endpoint; Test type: Superiority or Other; 95% exact binomial CI of proportion; Incidence Rate = 60, 95% CI [15 to 95]

2. Secondary Outcome: Participant Survival at 12 Months Post-Transplant
Time Frame: 12 months post-transplant
Population: Intent to Treat Sample participants not terminating prior to 12 months.
Measure: Number; unit: Participants
Arm/Group | Immunosuppression Withdrawal
Number analyzed (Participants) | 4
Participants | 4
Statistical Analysis 1: Comparison: Immunosuppression Withdrawal; Proportion with 95% exact binomial confidence interval; Test type: Superiority or Other; 95% exact binomial CI of proportion; Incidence Rate = 100, 95% CI [40 to 100]

3. Secondary Outcome: Acute Rejection at 12-Months
Description: Incidence of acute rejection[1] at 12 months post-transplant
  1. Diagnosis of acute rejection was made by renal (kidney) biopsy using the Banff 97 criteria. The Banff 97 diagnostic category for renal allograft biopsies is an international standardized histopathological classification. Acute rejection is defined by a renal biopsy demonstrating a Banff 97 classification of Grade IA or greater[2]
  2. Reference: Racusen LC, Solez K, Colvin RB et al,The Banff 97 working classification of renal allograft pathology. Kidney Int,55: 713-723, 1999
Time Frame: 12 months post-transplant
Population: Intent to Treat Sample
Measure: Number; unit: Participants
Arm/Group | Immunosuppression Withdrawal
Number analyzed (Participants) | 5
Participants | 4
Statistical Analysis 1: Comparison: Immunosuppression Withdrawal; Proportion with 95% exact binomial confidence interval; Test type: Superiority or Other; 95% exact binomial CI of proportion; Incidence rate = 80, 95% CI [28 to 99]

4. Secondary Outcome: Tolerance Induction
Description: Time from transplantation to initiation of sirolimus withdrawal.
Time Frame: 48 months
Population: Intent to treat sample that initiated sirolimus withdrawal
Measure: Number; unit: Days
Arm/Group | Immunosuppression Withdrawal
Number analyzed (Participants) | 1
Days | 391

5. Secondary Outcome: Renal Function as Measured by Glomerular Filtration Rate (GFR) at 24 Weeks
Description: GFR utilizing clearance of iothalamate.
  GFR is an index of level of kidney function. A higher value means better kidney function.
Time Frame: 24 weeks post-transplant
Population: Intent to Treat Sample
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Immunosuppression Withdrawal
Number analyzed (Participants) | 3
mL/min/1.73m^2 | 62.0 (8.5)

6. Secondary Outcome: Graft Survival at 12 Months Post-transplant
Time Frame: 12 months post-transplant
Population: Intent to treat sample participants not terminating prior to 12 months
Measure: Number; unit: Participants
Arm/Group | Immunosuppression Withdrawal
Number analyzed (Participants) | 4
Participants | 4
Statistical Analysis 1: Comparison: Immunosuppression Withdrawal; Proportion with 95% exact binomial confidence interval; Test type: Superiority or Other; 95% exact binomial CI of proportion; Incidence Rate = 100, 95% CI [40 to 100]

7. Secondary Outcome: Time From Transplant to Acute Rejection
Description: Time (days) from transplant to occurrence of acute rejection[1]
  1. Diagnosis of acute rejection was made by renal (kidney) biopsy using the Banff 97 criteria. The Banff 97 diagnostic category for renal allograft biopsies is an international standardized histopathological classification. Acute rejection is defined by a renal biopsy demonstrating a Banff 97 classification of Grade IA or greater[2]
  2. Reference: Racusen LC, Solez K, Colvin RB et al,The Banff 97 working classification of renal allograft pathology. Kidney Int,55: 713-723, 1999
Time Frame: Transplantation until rejection occurs (participants followed up to four years post-transplantation)
Population: Intent to treat sample participants with rejection
Measure: Median (Full Range); unit: Days
Arm/Group | Immunosuppression Withdrawal
Number analyzed (Participants) | 4
Days | 15 (95.4) [1 to 200]

8. Secondary Outcome: Proportion of Participants Requiring Antilymphocyte Therapy for Acute Rejection
Description: Proportion of participants who experienced acute rejection[1] requiring antilymphocyte therapy
  1. Diagnosis of acute rejection was made by renal (kidney) biopsy using the Banff 97 criteria. The Banff 97 diagnostic category for renal allograft biopsies is an international standardized histopathological classification. Acute rejection is defined by a renal biopsy demonstrating a Banff 97 classification of Grade IA or greater[2]
  2. Reference: Racusen LC, Solez K, Colvin RB et al,The Banff 97 working classification of renal allograft pathology. Kidney Int,55: 713-723, 1999
Time Frame: Participants followed from transplantation until completion of study (up to four years post-transplantation)
Population: Intent to Treat Sample
Measure: Number; unit: Participants
Arm/Group | Immunosuppression Withdrawal
Number analyzed (Participants) | 5
Participants | 0
Statistical Analysis 1: Comparison: Immunosuppression Withdrawal; Proportion with 95% exact binomial confidence interval; Test type: Superiority or Other; 95% exact binomial CI of proportion; Incidence Rate = 0, 95% CI [0 to 52.2]

9. Secondary Outcome: Proportion of Participants With Post-transplant Infections
Description: Proportion of participants who experienced infections post-transplant. Participants were checked for any type of opportunistic infection at all study visits post-transplantation (up to 4 years post-transplantation)
Time Frame: Participants followed from transplantation until completion of study (up to four years post-transplantation)
Population: Intent to Treat Sample
Measure: Number; unit: Participants
Arm/Group | Immunosuppression Withdrawal
Number analyzed (Participants) | 5
Participants | 4
Statistical Analysis 1: Comparison: Immunosuppression Withdrawal; Proportion with 95% exact binomial confidence interval; Test type: Superiority or Other; 95% exact binomial CI of proportion; Incidence Rate = 80, 95% CI [28 to 99]

10. Secondary Outcome: Proportion of Participants With Wound Complications
Time Frame: Start of study to end of study
Population: Intent to Treat Sample
Measure: Number; unit: Participants
Arm/Group | Immunosuppression Withdrawal
Number analyzed (Participants) | 5
Participants | 0
Statistical Analysis 1: Comparison: Immunosuppression Withdrawal; Proportion with 95% exact binomial confidence interval; Test type: Superiority or Other; 95% exact binomial CI of proportion; Incidence Rate = 0, 95% CI [0 to 52.2]

11. Secondary Outcome: Proportion of Participants With Malignancies
Time Frame: Participants followed from transplantation until completion of study (up to four years post-transplantation)
Population: Intent to Treat Sample
Measure: Number; unit: Participants
Arm/Group | Immunosuppression Withdrawal
Number analyzed (Participants) | 5
Participants | 0
Statistical Analysis 1: Comparison: Immunosuppression Withdrawal; Proportion with 95% exact binomial confidence interval; Test type: Superiority or Other; 95% exact binomial CI of proportion; Incidence Rate = 0, 95% CI [0 to 52.2]

12. Secondary Outcome: Proportion of Participants With a Sirolimus Associated Adverse Event
Time Frame: Participants followed from transplantation until completion of study (up to four years post-transplantation)
Population: Intent to Treat Sample
Measure: Number; unit: Participants
Arm/Group | Immunosuppression Withdrawal
Number analyzed (Participants) | 5
Participants | 5
Statistical Analysis 1: Comparison: Immunosuppression Withdrawal; Proportion with 95% exact binomial confidence interval; Test type: Superiority or Other; 95% exact binomial CI of proportion; Incidence Rate = 100, 95% CI [47.8 to 100]

13. Secondary Outcome: Proportion of Participants With Chronic Allograft Nephropathy
Time Frame: Participants followed from transplantation until completion of study (up to four years post-transplantation)
Population: Intent to Treat Sample
Measure: Number; unit: Participants
Arm/Group | Immunosuppression Withdrawal
Number analyzed (Participants) | 5
Participants | 0
Statistical Analysis 1: Comparison: Immunosuppression Withdrawal; Proportion with 95% exact binomial confidence interval; Test type: Superiority or Other; 95% exact binomial CI of proportion; Incidence Rate = 0, 95% CI [0 to 52.2]

14. Secondary Outcome: Proportion of Participants With Delayed Graft Function
Time Frame: Participants followed from transplantation until completion of study (up to four years post-transplantation)
Population: Intent to Treat Sample
Measure: Number; unit: Participants
Arm/Group | Immunosuppression Withdrawal
Number analyzed (Participants) | 5
Participants | 0
Statistical Analysis 1: Comparison: Immunosuppression Withdrawal; Proportion with 95% exact binomial confidence interval; Test type: Superiority or Other; 95% exact binomial CI of proportion; Incidence Rate = 0, 95% CI [0 to 52.2]

15. Secondary Outcome: Proportion of Participants With Post-transplant Diabetes Mellitus
Time Frame: Participants followed from transplantation until completion of study (up to four years post-transplantation)
Population: Intent to Treat Sample
Measure: Number; unit: Participants
Arm/Group | Immunosuppression Withdrawal
Number analyzed (Participants) | 5
Participants | 1
Statistical Analysis 1: Comparison: Immunosuppression Withdrawal; Proportion with 95% exact binomial confidence interval; Test type: Superiority or Other; 95% exact binomial CI of proportion; Incidence Rate = 20, 95% CI [0.5 to 71.6]

ADVERSE EVENTS:
Arm/Group | Immunosuppression Withdrawal
Serious Adverse Events (participants affected / at risk) | 4/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunosuppression Withdrawal (N=5)
Lymphocele (Blood and lymphatic system disorders) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 4 (5)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunosuppression Withdrawal (N=5)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 2 (3)
Thrombocythaemia (Blood and lymphatic system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Mouth ulceration (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (5)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (4)
Malaise (General disorders) | 1 (1)
Oedema (General disorders) | 3 (4)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
BK virus infection (Infections and infestations) | 2 (2)
Cytomegalovirus viraemia (Infections and infestations) | 1 (3)
Diverticulitis (Infections and infestations) | 1 (1)
Epstein-Barr viraemia (Infections and infestations) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Herpes virus infection (Infections and infestations) | 1 (4)
Oral infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1)
Graft dysfunction (Injury, poisoning and procedural complications) | 1 (2)
Incision site pain (Injury, poisoning and procedural complications) | 2 (2)
Medical device pain (Injury, poisoning and procedural complications) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (2)
Blood creatinine increased (Investigations) | 1 (1)
Weight increased (Investigations) | 2 (3)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Headache (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (2)
Dysuria (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal disorder (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Scrotal oedema (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial was stopped early due to meeting an acute rejection threshold of three acute rejections based on local pathology reads in the first five participants enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No